CLINICAL TRIAL: NCT03177655
Title: Effect of Guided Imagery on Well-being in Patients With Multiple Sclerosis
Acronym: HLGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Paul J. Mills, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121412
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Imagery (Experimental): Guided Imagery meditation
  Interventions: Other: Guided Imagery
- Journaling (Active Comparator): Keeping a journal
  Interventions: Other: Journaling

INTERVENTIONS:
Other: Guided Imagery — Guided Imagery meditation
  Arms: Guided Imagery
Other: Journaling — Keeping a journal
  Arms: Journaling

SUMMARY:
This single-center interventional study quasi-randomly allocated patients to a guided imagery or control intervention (positive journaling). Data were analyzed with treatment allocation masked.

DETAILED DESCRIPTION:
Interventions: Participants were assigned in alternate order to 10 weekly 1-hour sessions "Healing Light Guided Imagery" or at-home positive journaling; drop-outs were replaced.

Intervention Type: Behavioral

Multiple sclerosis (MS) is an autoimmune disease that affects the brain and spinal cord (central nervous system). Because nerves in any part of the brain or spinal cord may be damaged, patients with multiple sclerosis can have symptoms in different parts of the body. Many Multiple Sclerosis patients suffer from depression, fatigue and anxiety in addition to physical symptoms. Drugs prescribed for MS have been shown to not improve these comorbid psychological symptoms. Researchers have shown that mindfulness-based training programs can help MS patients, but these therapies are highly resource demanding and taxing for those involved. "Healing Light" Guided Imagery (HLGI; supplementary materials) is a guided imagery therapy that simulates a self-hypnotic trance state that has been anecdotally shown to improve depression and fatigue in patients with MS in less time and with fewer support resources. The investigators plan to test whether HLGI can increase patient well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Relapsing-Remitting Multiple Sclerosis
2. 18-70 years old
3. Able to read and write in English
4. Able to attend sessions at the UC San Diego School of Medicine

   * Age group: adult
   * Gender: both
   * Target enrollment: 20

Participant exclusion criteria:

1. Severe depression (score of 31 or higher on the BDI)
2. Very high levels of fatigue (above an average of 6 on the FSS)
3. Low levels of mindfulness (below an average score of 2 on the FMI).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life (MS-QOL-54) | Change from baseline at 10 weeks
  Quality of Life based on Multiple Sclerosis Quality of Life Instrument (MS-QOL-54)

SECONDARY OUTCOMES:
Mood (BDI-II) | Change from baseline at 10 weeks
  Depressed mood based on the Beck Depression Inventory II (BDI-II)
Fatigue (FSS) | Change from baseline at 10 weeks
  Fatigue levels based on the Fatigue Severity Scale (FSS)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided